CLINICAL TRIAL: NCT04432363
Title: Effects of Transcranial Direct Current Stimulation on Primary Cortex and Prefrontal Dorsolateral Cortex in Pain Processing on Healthy Volunteers: A Triple Blind Randomized Controlled Trial.
Brief Title: Effects of tDCS in M1 and DLPFC on Pain Processing in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Associate Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30012020204820
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Pain Processing in Healthy Volunteers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Three groups cross over study with two intervention groups and one sham group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M1 stimulation (Active Comparator): A 20 minutes 1mA direct current stimulation over left M1.
  Interventions: Device: Transcranial direct current stimulation
- M1+DLPFC stimulation (Active Comparator): A 20 minutes 1mA direct current stimulation over left M1 and 1mA direct current stimulation over left DLPFC.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): A 20 minutes sham stimulation where the device only is working first 30s and last 30s of the intervention and have a 10 seconds fade out in intensity at each ramp.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Direct current application over the scalp to stimulate and change the excitability of the cortical areas underneath the electrodes (in this case left primary motor cortex and left dorsolateral prefrontal cortex).

SUMMARY:
The purpose of this study is to evaluate the effects of a direct current applied transcranial over two cortical areas on healthy volunteers' pain processing.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Comprehension of the study tasks

Exclusion Criteria:

* Presence of pain in the previous 6 months
* Altered sensitivity in the tested regions
* Intolerance to electrotherapy
* Presence of pacemakers or any other implanted device
* Ulcers or scars in the skin at the location of the electrodes
* Treatment with direct current stimulation within one week
* Pregnancy
* Frequent headaches
* Epilepsy
* History of neuromuscular disease
* Previous clinical history of cervical surgery
* Injuries or surgery affecting the upper limb
* diabetes mellitus
* Cardiovascular diseases
* Oncological diseases
* Consumption of analgesic drugs 7 days before the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | Pre-intervention and immediately after treatment
  Pain pressure threshold change after a painful ischemic stimulus
Pain pressure algometer temporal summation | Pre-intervention and immediately after treatment
  Change in pain perceived between the first and tenth painful pressure stimulus

SECONDARY OUTCOMES:
Pain pressure threshold | Pre-intervention and immediately after treatment
  Measurement of pressure applied until the perception of pain
Pain pressure tolerance | Pre-intervention and immediately after treatment
  Measurement of maximal painful pressure tolerate using a pressure algometer
Neural mechanosensitivity | Pre-intervention and immediately after treatment
  Measurement of range of motion achieved until the perception of tension
Cold hyperalgesia with a cold pack | Pre-intervention and immediately after treatment
  Pain rated in a visual analogue scale after 10 seconds of a cold stimulus
Isometric grip strength | Pre-intervention and immediately after treatment
  Maximal pressure achieved in a isometric gripping task

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernandez Carnero, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rey Juan Carlos University — http://www.urjc.es